CLINICAL TRIAL: NCT05936021
Title: Clinical Validation Study for Optimization of Anemia MAnagement in Hemodialysis Patients With End Stage Kidney Disease Using the Dialysis Anemia TReatmenT Model
Acronym: SMART
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: SMART Study
Record Dates: First submitted 2023-06-27; First posted 2023-07-07 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Dialysis
Keywords: darbepoetin; kidney; dialysis; hemoglobin cycling
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: All patients placed on dialysis receive standard of care for a minimum of 150 days; after qualifying for the study, they enter the experimental intervention arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (Other): All patients placed on dialysis receive standard of care
  Interventions: Procedure: Standard of care
- Model-based Aranesp doses (Experimental): On entering the study cohort, patients will begin receiving doses calculated by the algorithm instead of by the standard of care procedures. Model-based Aranesp doses will be computed at the same time that doses based on the dialysis anemia protocol are determined. The model-based doses will be administered instead of the protocol-based doses and in the same way and at the same time as the protocol-based doses would have been.
  Interventions: Procedure: Algorithm model-based Aranesp doses

INTERVENTIONS:
Procedure: Algorithm model-based Aranesp doses — Patients will receive doses calculated by the algorithm instead of by the standard of care procedures. Model-based Aranesp doses will be computed at the same time that doses based on the dialysis anemia protocol are determined. The model-based doses will be administered instead of the protocol-based doses and in the same way and at the same time as the protocol-based doses would have been. The model-based dosing will be more flexible than the protocol-based dosing. Some constraints in the protocol-based dosing were created to prevent patients from achieving high Hb levels. The model-based dosing will also prevent these high Hb values but will do so by predicting a patient's Hb level into the future and then using these predictions to determine doses to reduce Hb variability and to reduce the amount of Aranesp used.
  Arms: Model-based Aranesp doses
Procedure: Standard of care — Current standard of care guidelines are followed for erythropoiesis-stimulating agents to control anemia in dialysis patients
  Arms: Standard of care

SUMMARY:
This is a human subject research study conducted in patients undergoing dialysis treatment with darbepoetin alfa at Intermountain Utah Dialysis and Intermountain Medical Center Dialysis Services. The purpose is to test a dose recommendation algorithm that may reduce hemoglobin variability and drug cost.

DETAILED DESCRIPTION:
Hemoglobin cycling is an outcome of treating long-term dialysis patients for anemia using erythropoiesis-stimulating agents (ESAs), and represents a conundrum for practitioners. While patients with low hemoglobin levels suffer from anemia, high hemoglobin levels may lead to blood clots and subsequent health risks. The current protocol for ESA dosing often results in suboptimal dosing that leads to hemoglobin cycling, which can have a negative impact on patient survival. To this end, we have developed a personalized method for ESA dosing that controls anemia in dialysis patients that is similar to the commercial product sold by PhySoft. Our method, the Dialysis Anemia Treatment Model, uses a mathematical model for erythropoiesis that takes each patient's physiology into account, predicting the optimal dose of ESA for that patient to prevent hemoglobin cycling. The goal of this computer-aided approach is to reduce hemoglobin cycling and the amount of drug used by predicting optimal doses to keep the patient's hemoglobin within the desired range. This is a human subject research study to validate the model in the clinic and demonstrate that it is able to minimize hemoglobin cycling in patients and reduce the amount of ESA drug administered.

ELIGIBILITY:
Inclusion Criteria:

* Males and females (≥ 18 years of age) with End Stage Kidney Disease undergoing in-center hemodialysis
* 150 days of hemoglobin readings and Aranesp doses without a hospitalization relevant to the condition of anemia

Exclusion Criteria:

* Inflammation as characterized by ferritin levels greater than 1000 ng/mL
* Patients with active cancer
* Patients with PTH greater than 1,000 pg/mL
* Active GI Bleed
* Hospitalization relevant to ESRD in last 150 days or during study
* Patients receiving Procrit rather than Aranesp.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Reduction of hemoglobin cycling in dialysis patients | 90 days after the intervention
  Reduction of hemoglobin cycling
Time hemoglobin levels are maintained within acceptable range | 90 days after the intervention
  Time hemoglobin levels are maintained within acceptable range

SECONDARY OUTCOMES:
Reduction in quantity of drug administered to patients | 90 days after the intervention
  Reduction in quantity of drug administered to patients

CONTACTS AND LOCATIONS:
Overall Officials: Chemiti Gopal, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (2):
- United States (2):
  - Intermountain Kidney Clinic, Murray, Utah
  - Dialysis Services, Murray, Utah